CLINICAL TRIAL: NCT03533829
Title: Preventing Post-Vaccination Presyncope and Syncope in Adolescents Using Simple, Clinic-based Interventions: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: PRO00094074; 200 2012 53663 0013 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Syncope, Vasovagal
Keywords: vaccination; pre-syncope; syncope prevention
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Buzzy® (Active Comparator): Buzzy® Drug Free Pain Relief which is a medical device designed to reduce vaccination pain when applied to the arm prior to and during a vaccination.
  Interventions: Device: Buzzy®
- Music (Active Comparator): Music will be selected and listened to as a distraction before and during vaccination.
  Interventions: Behavioral: Music
- Buzzy® and Music (Active Comparator): Buzzy® will be applied to the arm prior to and during vaccination and music will be selected and listened to before and during vaccination.
  Interventions: Device: Buzzy®; Behavioral: Music

INTERVENTIONS:
Device: Buzzy® — Buzzy® Drug Free Pain Relief which is a medical device designed to reduce vaccination pain when applied to the arm prior to and during a vaccination.
  Arms: Buzzy®; Buzzy® and Music
Behavioral: Music — Music will be selected and listened to as a distraction before and during vaccination.
  Arms: Buzzy® and Music; Music

SUMMARY:
This is a randomized controlled open-label trial. During the study, adolescents scheduled to receive at least one intramuscular (IM) vaccine will receive either Buzzy®, Music, or Buzzy® and Music intervention(s) in addition to standard care to evaluate the feasibility and acceptability of these interventions prior to being used in a larger study to assess the effectiveness of the interventions in preventing post-vaccination presyncope and syncope. Feasibility will be assessed according to study staff ability to successfully administer the protocol specified clinic-based interventions and per both study staff and healthcare provider responses to written feasibility assessments. Acceptability will be assessed according to the participant's self-report. In addition, baseline needle phobia and anxiety, post-vaccination pain and presyncope symptoms, and pre- and post- vaccination state anxiety will be assessed per participant written self-report to standardized survey questions.

ELIGIBILITY:
Inclusion Criteria:

1. 10 years through 17 years of age
2. If 10 through 13 years of age, the subject must be receiving at least one vaccine delivered intramuscularly
3. If 14 through 17 years of age, the subject must be receiving at least two injectable vaccines one of which must be delivered intramuscularly
4. The parent/guardian must be willing and capable of providing written informed consent for the adolescent and the adolescent must be willing and capable of providing assent.
5. The subject must be willing to stay for the completion of all study-related activities.
6. Parent/guardian and adolescent must speak and read English by self-report

Exclusion Criteria:

1. Receipt of investigational or experimental vaccine or medication within the previous two weeks
2. Receipt of routine injectable medication
3. Permanent indwelling venous catheter
4. Blood drawn within the past hour or scheduled for a blood draw during the post-vaccination observation period
5. Injection of medication during the past hour or scheduled for injection of medication during the observation period.
6. Cold intolerance or cold urticaria
7. Raynaud's phenomenon
8. Sickle cell disease
9. Inability to hear
10. Significant visual impairment or blindness
11. Febrile or acutely ill individuals
12. Upper arm or shoulder pain or injury
13. Adolescent or parent/Guardian is an immediate relative of study staff or an employee who is supervised by study staff.
14. Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel "Chip" B Walter, MD, MPH, Principal Investigator — Duke Univeristy; Theresa Harrington, MD, MPH&TM, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buzzy® | Music | Buzzy® and Music
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adolescents randomized to intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Buzzy® | Music | Buzzy® and Music | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Count of Participants; unit: Participants]
  10-13 years | 8 | 6 | 10 | 24
  14-17 years | 2 | 4 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 7 | 7 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 2 | 2 | 2 | 6
  Race: White | 7 | 8 | 7 | 22
  Race: More than one race | 0 | 0 | 1 | 1
  Race: Other race | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Have Buzzy® Applied to and Kept at Vaccination Site/s for ≥ 30 Seconds Prior to Vaccination
Description: Buzzy® will be applied to and kept on the subjects arm for a minimum of 30 seconds prior to vaccination.
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 10 | 0 | 10

2. Primary Outcome: Number of Subjects Who Have Buzzy® Kept on Vaccination Arm/s During the Entire Vaccination Procedure
Description: Buzzy® will be applied to and kept on the subjects arm for the duration of the vaccination procedure.
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 9 | 0 | 10

3. Primary Outcome: Number of Subjects Who Have Music Playing for ≥ 3 Minutes Prior to Vaccination
Description: Music will be played over speakers for a minimum of 3 minutes prior to vaccination
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 10 | 10

4. Primary Outcome: Number of Subjects Who Have Music Playing for 10 Minutes Post Vaccination
Description: Music will be played over speakers through the 10 minute post vaccination pain assessment
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 8 | 7

5. Primary Outcome: Number of Subjects Who Complete the Pre-vaccination Anxiety Assessment
Description: Subjects will be asked to complete an anxiety assessment prior to vaccination
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

6. Primary Outcome: Number of Subjects Who Complete the Pre-vaccination Needle Phobia Assessment
Description: Subjects will be asked to complete a needle phobia assessment pre-vaccination
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

7. Primary Outcome: Number of Subjects Who Complete the Post-vaccination Pain Assessment at 1 Minute.
Description: Subjects will complete a post vaccination pain assessment within one minute of their final vaccination
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 4 | 7 | 3

8. Primary Outcome: Number of Subjects Who Complete the Post-vaccination Pain Assessment at 10 Minutes
Description: Subjects will complete a post vaccination pain assessment at 10 minutes after their final vaccination
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 8 | 10 | 9

9. Primary Outcome: Number of Subjects Who Complete the Post-vaccination Presyncope Symptom Assessment
Description: Subjects will complete a questionnaire about presyncope symptoms after their vaccination/s
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

10. Primary Outcome: Number of Subjects Who Complete the Post Vaccination Anxiety Assessment
Description: Subjects will complete a post vaccination anxiety assessment
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

11. Primary Outcome: Number of Subjects Who Complete the Acceptability Assessment
Description: Subjects will be given a questionnaire about the acceptability of their intervention.
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

12. Primary Outcome: Number of Reports From Coordinators That Indicated Having Music Playing During the Vaccine Administration Was Somewhat Easy or Very Easy
Description: Coordinators will answer a questionnaire about the feasibility of the music intervention after each encounter with a subject
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 5 | 6

13. Primary Outcome: Number of Reports From Coordinators That Indicated Having Music Playing During the Vaccine Administration Was Somewhat Assistive or Very Assistive
Description: as for outcome 12
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 4 | 3

14. Primary Outcome: Number of Reports From Coordinators That Indicated Having Buzzy® Applied in Conjunction With the Vaccination Was Somewhat Easy or Very Easy
Description: Coordinators will answer a questionnaire about the feasibility of the Buzzy® intervention after each encounter with a subject
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 9 | 0 | 6

15. Primary Outcome: Number of Reports From Coordinators That Indicated Having Buzzy® Applied in Conjunction With the Vaccination Was Somewhat Assistive or Very Assistive
Description: as for outcome 14
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 9 | 0 | 5

16. Primary Outcome: Number of Reports From Providers That Indicated Having Music Playing During the Vaccine Administration Was Somewhat Easy or Very Easy
Description: Providers will answer a questionnaire about the feasibility of the music intervention after each encounter with a subject
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated. One participant did not complete the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 9
Participants | 0 | 7 | 8

17. Primary Outcome: Number of Reports From Providers That Indicated Having Music Playing During the Vaccine Administration Was Somewhat Assistive or Very Assistive
Description: as for outcome 16
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated. One participant did not complete the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 9
Participants | 0 | 6 | 7

18. Primary Outcome: Number of Reports From Providers That Indicated Having Buzzy® Applied in Conjunction With the Vaccination Was Somewhat Easy or Very Easy
Description: Providers will answer a questionnaire about the feasibility of the Buzzy® intervention after each encounter with a subject
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated. One participant did not complete the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 9 | 0 | 10
Participants | 6 | 0 | 8

19. Primary Outcome: Number of Reports From Providers That Indicated Having Buzzy® Applied in Conjunction With the Vaccination Was Somewhat Assistive or Very Assistive
Description: as for outcome 18
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 7 | 0 | 7

20. Primary Outcome: Number of Subjects Who Like Having Music Play During Their Shot/s a Little or Very Much
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 9 | 9

21. Primary Outcome: Number of Subjects Who Felt Having Music Play During Their Shot/s Was Somewhat Easy or Easy
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 9 | 10

22. Primary Outcome: Number of Subjects Who Found Music Playing While Receiving Their Shots to be Somewhat Comfortable or Very Comfortable
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated. One participant did not complete the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 9
Participants | 0 | 10 | 9

23. Primary Outcome: Number of Subjects Who Found the Music Playing While They Got Their Shot/s to be Just Right
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 10 | 8

24. Primary Outcome: Number of Subjects Who Would be Somewhat Likely or Very Likely to Want to Listen to Music Again While Receiving Shot/s
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 10 | 10

25. Primary Outcome: Number of Subjects Who Found the Music App Sufficient or Somewhat Sufficient to Selecting the Music They Like
Description: Subjects will complete a survey about the acceptability of the music intervention during their vaccinations
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 0 | 10 | 10
Participants | 0 | 10 | 10

26. Primary Outcome: Number of Subjects Who Either Like a Little or Very Much Liked Having Buzzy® on Their Arm/s During Shot/s
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 9 | 0 | 9

27. Primary Outcome: Number of Subjects Who Found Having Buzzy® on Their Arm/s During Shot/s Somewhat Easy or Very Easy
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participant randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 10 | 0 | 9

28. Primary Outcome: Number of Subjects Who Found Having Buzzy® on Their Arm/s During Shot/s Somewhat Comfortable or Very Comfortable
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 7 | 0 | 8

29. Primary Outcome: Number of Subjects Who Were Not Bothered by the Cold Temperature of Buzzy® on Their Arm/s During Shot/s
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 6 | 0 | 8

30. Primary Outcome: Number of Subjects Who Were Not Bothered by the Vibration of Buzzy® on Their Arm/s During Shot/s
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 10 | 0 | 9

31. Primary Outcome: Number of Subjects Who Would Choose to Have Buzzy® on Their Arm/s During Shot/s Again
Description: Subjects will complete a survey about the acceptability of the Buzzy® intervention during their vaccinations
Time Frame: Day1
Population: Participants randomized to intervention and vaccinated
Measure: Count of Participants; unit: Participants
Arm/Group | Buzzy® | Music | Buzzy® and Music
Number analyzed (Participants) | 10 | 0 | 10
Participants | 9 | 0 | 8

ADVERSE EVENTS:
Time Frame: Data were collected for 20 minutes post-vaccination.
Arm/Group | Buzzy® | Music | Buzzy® and Music
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buzzy® (N=10) | Music (N=10) | Buzzy® and Music (N=10)
Presyncope (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Air conditioning in room not working. The patient felt better after being fanned for five minutes. Symptoms lasted between 1 and 5 minutes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03533829/Prot_SAP_000.pdf